CLINICAL TRIAL: NCT06284616
Title: Benefits of a Juvenile Arthritis Support Program (JASP-1) for Children Recently Diagnosed With Juvenile Idiopathic Arthritis (JIA) and Their Parents
Brief Title: JASP-1 for Children Recently Diagnosed and Their Parents
Acronym: JASP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K2019-0392
Record Dates: First submitted 2024-02-13; First posted 2024-02-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: JIA; Support Program; Patient Satisfaction; Patient Outcome Assessment
Keywords: JIA; Support program; Patient Satisfaction; Patient outcome assessment
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The study is a non-randomized intervention study with 2 groups receiving either a Support program (JASP-1) or standard care
Masking Description: All patient receiving a JIA diagnose was offered to participate in JASP-1. The controls had received diagnose before the start of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JASP-1 group (Experimental): Participants were recruited from August 2019 to April 2022. The JASP-1 group consisted of children 0-16 years old who were diagnosed with JIA at their first visit to the PRC and their parents
  Interventions: Behavioral: JASP-1
- Control group (No Intervention): The control group consisted of children 1-16 years old, who were diagnosed with JIA at their first visit at the PRC who were receiving standard care after the diagnosis, and their parents

INTERVENTIONS:
Behavioral: JASP-1 — patients following the Juvenile Arthritis Support Program at the Pediatric Rheumatology Clinic
  Arms: JASP-1 group

SUMMARY:
To implement and evaluate a patient-and family-centered Juvenile Arthritis Support Program during one year (JASP-1) for children recently diagnosed with JIA and their parents and after 12 months compare satistaction with care and health outcomes with a control group receiving standard care.

DETAILED DESCRIPTION:
Children diagnosed with JIA (n=50) and their parents were offered the opportunity to participate in the JASP-1 from the time of diagnosis and the following year. One year after the JIA diagnosis, the children and/or their parents were invited to answer a study-specific questionnaire comprising 16 questions. The questionnaire assessed their experiences with the information, communication, participation, and emotional support they had received during the first year with JIA. In order to compare outcomes, the questionnaire was answered by both participants in JASP-1 and patients and parents receiving standard care (n=25).

One example of a question is; If you asked questions to the health care professionals, did you get answers that you understood? Response alternatives range from "No, not at all" to "Yes, Completely" ona 5-point Likert scale.

In Swedish Pediatric Rheumatology Quality Register (PedSRQ) information about treatment, disease- and joint activity (registered by Medical doctor), and Patient Reported Outcome Measures (PROM), are measured. The total Child Health Activity Questionnaire (CHAQ-score), as well as active joints and treatment at 12 months was registered in the PedSRQ and analyzed.

The study specific questionnaire measuring patient satisfaction has been developed in collaboration with the Swedish Municipalities and County councils.

Experimental and descriptive analyses will be performed using software for statistical analysis, SPSS. Distributions of responses will be calculated in percentage. Differences in proportions between groups will be determined by performing chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-16 years old
* Diagnosed with JIA at their first visit to the PRC

Exclusion Criteria:

* Children that did not fulfil the criteria for JIA
* Children/parents who could not understand the Swedish language.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of Patient Reported Experienced Measures (PREM) | 12 months
  A study specific PREM questionnaire with 16 items. 5 point likert scale

SECONDARY OUTCOMES:
Rate of Overall perceived health | 12 months
  One item on a 5 point likert scale, range from "not good at all" to "totally good"
Rate of Child Health Activity Questionnaire (CHAQ) | 12 months
  CHAQ assesses functional ability and assists in understanding the impact of the disease on the child´s daily life. On a Visual Analog Scale (VAS) ranging 0 to 10
Number of active joints | 12 months
  Medical doctors assessment of the childs actice joints

CONTACTS AND LOCATIONS:
Overall Officials: Eva Broström, Professor, Principal Investigator — Supervisor
Locations (1):
- Astrid Lindgren Children´s Hospital, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mordrup K, Jungner JG, Brostrom E, Palmblad K, Bartholdson C. Benefits of a Juvenile Arthritis Support Program (JASP-1) for children recently diagnosed with Juvenile Idiopathic Arthritis and their parents. BMC Rheumatol. 2024 Aug 15;8(1):35. doi: 10.1186/s41927-024-00404-8. PMID 39143588